CLINICAL TRIAL: NCT02183597
Title: Whole-body MRI for the Detection of Metastasis
Acronym: WBMRI
Status: Withdrawn | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: STUC-2013-WBMRI-Sitter
Record Dates: First submitted 2014-05-16; First posted 2014-07-08 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer; Metastases
Keywords: Magnetic Resonance Imaging; Data Accuracy; Reproducibility of Results; Diagnosis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced breast cancer: Women with advanced breast cancer

SUMMARY:
Develop and optimize protocols for whole body MRI for detection of metastases. Evaluate diagnostic accuracy through application of optimized protocols for screening of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

- Cancer patient

Exclusion Criteria:

* Poor general condition
* Pacemaker or other MRI contraindications

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in Mid Norway living with advanced breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of metastasis in skeleton | Baseline and after 6 months
  Number of skeleton metastasis will be assessed at the regular clinical follow-up of breast cancer patients with metastatic disease

CONTACTS AND LOCATIONS:
Overall Officials: Beathe Sitter, PhD, Principal Investigator — Norwegian University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided